CLINICAL TRIAL: NCT00717496
Title: Telephone Support Intervention to Improve Breastfeeding Rates in Low-Income Women
Brief Title: Telephone Support Intervention to Improve Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 04-0893; 04-0893
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2008-07

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Telephone Support; Latino
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The intervention will consist of outreach telephone calls daily by bilingual trained nursing staff for the first 2 weeks postpartum using the scripted protocols developed for this program. This group will receive a small bag with reading materials, illustrations of breastfeeding positions and latch, hand breast pump, and lanolin cream. The intervention nurse will ask the mothers on their initial intake call for the best time to call each day to minimize time needed to reach the mother.
  Interventions: Other: Telephone Support Intervention to Improve Breastfeeding
- B (No Intervention): Mothers assigned to the control group will receive usual care. This group will also receive a small bag with reading materials, illustrations of breastfeeding positions and latch, hand breast pump, and lanolin cream.

INTERVENTIONS:
Other: Telephone Support Intervention to Improve Breastfeeding — The intervention will consist of outreach telephone calls daily by bilingual trained nursing staff for the first 2 weeks postpartum using the scripted protocols developed for this program. Both groups will receive a small bag with reading materials, illustrations of breastfeeding positions and latch, hand breast pump, and lanolin cream. The intervention nurse will ask the mothers on their initial intake call for the best time to call each day to minimize time needed to reach the mother.
  Arms: A

SUMMARY:
This randomized controlled trial will evaluate an innovative telephone-based breastfeeding education and promotion intervention that will be implemented in a low-income, predominately Latina population. The trial will assess the impact of the intervention on duration of breastfeeding and exclusivity of breastfeeding at 1, 2, 3 and 6 months post-partum.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate an innovative telephone-based breastfeeding education and promotion intervention that will be implemented in a low-income, predominately Latina population. The intervention was developed in association with national breastfeeding experts, local public health department and WIC personnel and community leaders. Additionally, it will also be informed by focus groups that are currently being conducted in the community with a particular emphasis on cultural barriers to breastfeeding in Latina populations. The intervention consists of scripted education and support protocols delivered by telephone daily, in English and Spanish, by a trained nurse over the first two weeks after delivery and will be funded by the Division of General Pediatrics. In the evaluation mothers will be randomized during the first 24 hours after delivering a healthy baby to the intervention arm or to usual post-partum care. The trial will assess the impact of the intervention on duration of breastfeeding and exclusivity of breastfeeding at 1, 2, 3 and 6 months post-partum. In addition, it will assess cost-effectiveness of the intervention and secondary and process-of-care outcomes related to maternal satisfaction with feeding, confidence with breastfeeding and utilization of health services.

The specific aims of this project are:

* To evaluate in a randomized controlled trial the effect of a telephone-based breastfeeding support and education intervention compared to usual post-partum care on a) the duration of breastfeeding at 1, 2, 3 and 6 months and b) the exclusivity of breastfeeding at 1, 2, 3 and 6 months in low-income, primarily Latina women.
* To evaluate the cost-effectiveness of the telephone-based intervention compared to usual care
* To compare secondary outcomes for mothers in the intervention versus control groups such as maternal satisfaction and confidence with feeding, reasons for discontinuing breastfeeding and utilization of acute, preventive health care services and hospitalizations
* To better understand unmet needs in women who breastfeed and how well the intervention addressed these needs by conducting qualitative interviews

The major hypotheses are:

1. a) Proactive telephone contact in the early postpartum period using scripted protocols will increase breastfeeding rates in low-income women from a current baseline of 30% to 45% at 3 months and from 20% to 35% at 6 months.

   b) Proactive telephone contact in the early postpartum period using scripted protocols will increase exclusivity from a current baseline of 15% at 3 months to 30% and from 10% at 6 months to 25% compared to the usual care group.
2. The telephone-based intervention will be cost-effective compared with routine care with use of formula.
3. The telephone-based intervention will be associated with higher levels of maternal satisfaction overall.
4. Confidence with breastfeeding will be higher in breastfeeding mothers in the intervention group compared to breastfeeding mothers in the usual care group.
5. Compliance with scheduled preventive visits will be higher in the intervention group and use of acute health services, including clinic and emergency room visits will be lower in the intervention group compared to the usual care group. Hospitalizations will not differ significantly between the groups.

ELIGIBILITY:
Inclusion Criteria:

* First time mother
* Mother 18 years old or older
* 37 weeks gestation or greater at delivery
* Intent to breastfeed

Exclusion Criteria:

* mother's primary language is something other than English or Spanish
* mother has medical complications that interfere with her instituting breastfeeding or require her to stay in the hospital for >72 hours
* infant has a medical problem that requires admission to the intensive care nursery or requires hospitalization for >72 hours
* mother expresses a strong desire to formula feed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Breastfeeding at 3 months and at 6 months | 3 months and six months

SECONDARY OUTCOMES:
Exclusively breastfeeding at 3 months and at 6 months | 3 months and 6 months
Cost analysis: costs of training, costs of nurse for intervention, costs associated with intervention, cost of formula from WIC, time spent breastfeeding and time spent getting formula, acute care utilization associated with breastfeeding problems | 6 months
Maternal satisfaction: 4-point Likert scale of satisfaction | 6 months
Maternal confidence among breastfeeding mothers: Breastfeeding Self-Efficacy Short Form, 14-item scale scored 1-5, with range of scores from 14-70 | 3 months and 6 months
Reasons for stopping breastfeeding-descriptive data | 6 months
Utilization outcomes: number of preventive care visits; number of acute visits for illness to clinic; number of emergency room visits; number of hospitalizations | 6 months
Descriptive data regarding problems encountered, unmet needs, areas of strength and weakness of intervention and ways it could be improved. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Breastfeeding and the use of human milk. American Academy of Pediatrics. Work Group on Breastfeeding. Pediatrics. 1997 Dec;100(6):1035-9. doi: 10.1542/peds.100.6.1035. PMID 9411381
- [Background] U.S. Department of Health and Human Services. Healthy People 2010. 2000:47-8.
- [Background] Zimmerman DR, Guttman N. "Breast is best": knowledge among low-income mothers is not enough. J Hum Lact. 2001 Feb;17(1):14-9. doi: 10.1177/089033440101700104. PMID 11847846
- [Background] Forste R, Weiss J, Lippincott E. The decision to breastfeed in the United States: does race matter? Pediatrics. 2001 Aug;108(2):291-6. doi: 10.1542/peds.108.2.291. PMID 11483790
- [Background] Li R, Grummer-Strawn L. Racial and ethnic disparities in breastfeeding among United States infants: Third National Health and Nutrition Examination Survey, 1988-1994. Birth. 2002 Dec;29(4):251-7. doi: 10.1046/j.1523-536x.2002.00199.x. PMID 12431264
- [Background] Loughlin HH, Clapp-Channing NE, Gehlbach SH, Pollard JC, McCutchen TM. Early termination of breast-feeding: identifying those at risk. Pediatrics. 1985 Mar;75(3):508-13. PMID 3975119
- [Background] Taveras EM, Capra AM, Braveman PA, Jensvold NG, Escobar GJ, Lieu TA. Clinician support and psychosocial risk factors associated with breastfeeding discontinuation. Pediatrics. 2003 Jul;112(1 Pt 1):108-15. doi: 10.1542/peds.112.1.108. PMID 12837875
- [Background] Libbus MK. Breastfeeding attitudes in a sample of Spanish-speaking Hispanic American women. J Hum Lact. 2000 Aug;16(3):216-20. doi: 10.1177/089033440001600306. PMID 11153155
- [Background] Milligan RA, Pugh LC, Bronner YL, Spatz DL, Brown LP. Breastfeeding duration among low income women. J Midwifery Womens Health. 2000 May-Jun;45(3):246-52. doi: 10.1016/s1526-9523(00)00018-0. PMID 10907334
- [Background] Wood SP, Sasonoff KM, Beal JA. Breast-feeding attitudes and practices of Latino women: a descriptive study. J Am Acad Nurse Pract. 1998 Jun;10(6):253-60. doi: 10.1111/j.1745-7599.1998.tb00502.x. No abstract available. PMID 9801560
- [Background] Guise JM, Palda V, Westhoff C, Chan BK, Helfand M, Lieu TA; U.S. Preventive Services Task Force. The effectiveness of primary care-based interventions to promote breastfeeding: systematic evidence review and meta-analysis for the US Preventive Services Task Force. Ann Fam Med. 2003 Jul-Aug;1(2):70-8. doi: 10.1370/afm.56. PMID 15040435
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Derived] Gavine A, Shinwell SC, Buchanan P, Farre A, Wade A, Lynn F, Marshall J, Cumming SE, Dare S, McFadden A. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2022 Oct 25;10(10):CD001141. doi: 10.1002/14651858.CD001141.pub6. PMID 36282618
- [Derived] Bunik M, Shobe P, O'Connor ME, Beaty B, Langendoerfer S, Crane L, Kempe A. Are 2 weeks of daily breastfeeding support insufficient to overcome the influences of formula? Acad Pediatr. 2010 Jan-Feb;10(1):21-8. doi: 10.1016/j.acap.2009.09.014. PMID 20129478